CLINICAL TRIAL: NCT06935292
Title: Comparative Study Between Oral Melatonin and Nebulized Dexmedetomidine Premedication on Attenuation of Hemodynamic Response to Direct Laryngoscopy and Tracheal Intubation in Hypertensive Patients: A Prospective Randomized Trial
Brief Title: Oral Melatonin VS Nebulized Dexmedetomidine Premedication on Attenuation of Hemodynamic Response to Direct Laryngoscopy and Tracheal Intubation in Hypertensive Patients
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Aya Gamal Abo Elfotoh Ismaeil, Resident of Anesthesia, Surgical Intensive Care and Pain Management, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 36264MS867/3/25
Record Dates: First submitted 2025-04-11; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Tracheal Intubation Morbidity; Laryngoscopy; Hemodynamic Response
Keywords: Direct laryngoscope; Dexmedetomidine; Melatonin; Tracheal Intubation; Hypertension; Hemodynamic response
MeSH Terms: conditions — Hypertension | interventions — Dexmedetomidine; Melatonin

STUDY DESIGN:
Intervention Model Description: Dexmedetomidine will be given in the form of nebulized dexmedetomidine (1μg/kg) one hour before induction of anesthesia.
  Melatonin will be given as melatonin oral tablet (5mg) one hour before induction of anesthesia.
Who Masked: Investigator, Outcomes Assessor
Masking Description: A Research nurse who will not participate in the evaluation of sedation will give the drugs to all patients 60 minute before induction of general anesthesia. Outcome assessment will be conducted by an anesthesiologist who will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dexmedetomidine group (Experimental): Participants in this group will receive nebulized dexmedetomidine (1μg/kg) one hour before induction of anesthesia
  Interventions: Drug: Dexmedetomidine
- Melatonin group (Experimental): Participants in this group will receive melatonin oral tablet (5mg) one hour before induction of anesthesia
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Dexmedetomidine — Nebulized Dexmedetomidine (1μg/kg)
  Other Names: Precedex
  Arms: Dexmedetomidine group
Drug: Melatonin — Oral Melatonin tablet (5mg)
  Other Names: Circadin
  Arms: Melatonin group

SUMMARY:
The aim of this study is to compare the efficacy of oral melatonin versus nebulized dexmedetomidine in attenuating the hemodynamic response to direct laryngoscopy and endotracheal intubation in controlled hypertensive patients prepared for general anesthesia

DETAILED DESCRIPTION:
Laryngoscopy and endotracheal intubation are associated with sympathetic stimulation and induce hemodynamic changes with consequent increase in heart rate (HR) and blood pressure (BP) which may lead to myocardial infarction, cardiac arrhythmias, cardiac failure and cerebrovascular accidents in patients with underlying cardiovascular or cerebrovascular diseases.

Dexmedetomidine is a centrally acting α-2 adrenergic agonist with sedative, hypnotic, analgesic, anxiolytic, anti-sialagogue, antinociceptive and sympatholytic action. Premedication with dexmedetomidine through intravenous, intramuscular and intranasal route has been shown to effectively attenuate hemodynamic response to laryngoscopy and endotracheal intubation. Nebulization provides an alternative route of dexmedetomidine premedication with high bioavailability through both nasal (65%) and oral mucosa (82%) and avoids a venipuncture as a prerequisite. Recent studies have shown nebulization as a novel route of dexmedetomidine administration for attenuation of hemodynamic response to endotracheal intubation.

Melatonin is a natural substance produced mainly in the pineal gland of all mammals and vertebrates. It is rapidly distributed and eliminated after intravenous administration. After oral administration, plasma concentration peaks after 60 min and is then eliminated. It exerts its hypnotic effects through the activation of the Melatonin receptors type I and II (MT1, MT2). It has shown potent analgesic effects in a dose dependent manner in experimental studies. It may induce relaxation of the arterial wall smooth muscle by increasing nitric oxide levels. Therefore, premedication with sublingual/oral Melatonin is associated with pre-operative anxiolysis and sedation without impairment of orientation, psychomotor skills, or impact on quality of recovery, moreover, it attenuates the hemodynamic stress response to laryngoscopy and tracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Age (40-60) years of both genders.
* Controlled hypertensive patients.
* Categorized as ASA physical status II.
* Planning to do an elective surgery under General Anesthesia.

Exclusion Criteria:

* Patient refusal to participate in the study.
* Patient with expected difficult intubation.
* Body Mass Index (BMI) > 30 kg/m2.
* History of allergy to the drugs of the study.
* Patients with Heart rate<50 or Heart block.
* End stage renal and hepatic disease.
* Patients on beta blocker, oral hypoglycemics, anti-depressants, anti-convulsants, anti- psychotics and thyroid medications.
* Pregnant or lactating females.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Heart Rate (HR) | Till the end of surgery (up to 2 hours)
  Heart Rate will be assessed using pulse oximeter in pre-operative room (baseline), before the induction of anesthesia, immediately before laryngescopy or intubation, 1 minute after induction, 3 minutes after induction, 5 minutes after induction, every 30 minutes till the end of operation.

SECONDARY OUTCOMES:
Change in Systolic and Diastolic blood pressure | Till the end of surgery (up to 2 hours)
  Systolic and diastolic blood pressure will be recorded in pre-operative room (baseline), before the induction of anesthesia, immediately before laryngescopy or intubation, 1 minute after induction, 3 minutes after induction, 5 minutes after induction, every 30 minutes till the end of operation.
Sedation levels using Ramsay Sedation Scale | Till 2 hours after the surgery
  Sedation levels will be assessed using Ramsay Sedation Scale (1, Anxious and agitated, restless, or both; 2, Cooperative, oriented, and calm; 3 Responsive to commands only; 4 Exhibiting brisk response to light glabellar tap or loud auditory stimulus; 5, Exhibiting a sluggish response to light glabellar tap or loud auditory stimulus; 6, Unresponsive) before administration of the study drugs, before induction of anesthesia (60 minutes after drug taken), every 30 minutes post operative till 2 hours after surgery.
Intraoperative requirement of fentanyl | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).

CONTACTS AND LOCATIONS:
Overall Officials: Aya GAE Ismaeil, MBBCH, Principal Investigator — Faculty of Medicine, Tanta University, Egypt
Locations (1):
- Tanta University Hospital, Tanta, El-Gharbia Govenorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author